CLINICAL TRIAL: NCT02804750
Title: Phase 2 Study of the Safety and Efficacy of CORT125134 in the Treatment of Endogenous Cushing's Syndrome
Brief Title: Study to Evaluate CORT125134 in Participants With Cushing's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-451
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's Syndrome; Cushing's Disease; Cushing's; Hypercortisolemia; Cushingoid; Type 2 Diabetes; Impaired Glucose Intolerance; Hypertension; Adrenal Corticotrophic Hormone (ACTH); Adrenocortical Carcinoma; Primary Pigmented Nodular Adrenal Disease (PPNAD); Moon Facies; Dorsocervical Fat Pad; Adrenal Adenoma; Adrenal Carcinoma; Adrenal Autonomy; Cortisol
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; ACTH Syndrome, Ectopic; Diabetes Mellitus, Type 2; Hypertension; Adrenocortical Carcinoma; Adrenal Cortex Neoplasms | interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Low-dose Group (Experimental): 100 mg/day for 4 weeks in Period 1, then 150 mg/day for 4 weeks in Period 2, then 200 mg/day for 4 weeks in Period 3. There was no washout between treatment periods. Period 3 was followed by a 4-week follow-up period. Per-protocol, Group 1 did not participate in treatment Period 4.
  Interventions: Drug: CORT125134
- Group 2: High-dose Group (Experimental): 250 mg/day for 4 weeks in Period 1, then 300 mg/day for 4 weeks in Period 2, then 350 mg/day for 4 weeks in Period 3, then 400 mg/day for 4 weeks in Period 4. There was no washout between treatment periods. Period 4 was followed by a 4-week follow-up period.
  Interventions: Drug: CORT125134

INTERVENTIONS:
Drug: CORT125134

SUMMARY:
Cushing's syndrome is a relatively rare disorder caused by prolonged exposure to high levels of the glucocorticoid hormone cortisol. Cushing's syndrome may result from elevated endogenous or exogenous sources of cortisol. Endogenous Cushing's syndrome resulting from cortisol overproduction by the adrenal glands is the subject of this protocol.

Patients with exogenous Cushing's syndrome, which develops as a side effect of chronic administration of high doses of glucocorticoids, were not eligible for enrollment in this study.

The purpose of this study was to evaluate the safety and efficacy of CORT125134 for treatment of endogenous Cushing's syndrome. The multicenter study was conducted in the United States and in Europe.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study with two dose groups, each with a two-step dose escalation, designed to evaluate the safety and efficacy of CORT125134 for the treatment of endogenous Cushing's syndrome. CORT125134 was administered orally once daily for 16 weeks with dose escalations occurring every 4 weeks.

Pharmacokinetics (PK) profiles were generated at every dose level. A data review committee reviewed PK and safety data and recommended the final plan for dose escalation in Group 2.

ELIGIBILITY:
Inclusion Criteria:

1. Has a confirmed diagnosis of endogenous Cushing's syndrome.
2. Requires medical treatment of hypercortisolemia.
3. Meets at least one of the following criteria:

   1. Has type 2 diabetes mellitus.
   2. Has impaired glucose tolerance.
   3. Has hypertension.

Exclusion Criteria:

1. Has non-endogenous source of hypercortisolemia
2. Has uncontrolled, clinically significant hypothyroidism or hyperthyroidism
3. Has poorly controlled hypertension
4. Has Stage ≥ 4 renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas G Moraitis, MD, Study Director — Corcept Therapeutics
Locations (25):
- United States (12):
  - Laguna Hills, California
  - Aurora, Colorado
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Indianapolis, Indiana
  - Covington, Kentucky
  - Rochester, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Richmond, Virginia
- Hungary (2):
  - Budapest
  - Pécs
- Italy (8):
  - Cuneo
  - Messina
  - Milan
  - Naples
  - Orbassano
  - Roma
  - Siena
  - Torino
- Netherlands (2):
  - Leiden
  - Rotterdam
- Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivonello R, Munster PN, Terzolo M, Ferrigno R, Simeoli C, Puglisi S, Bali U, Moraitis AG. Glucocorticoid Receptor Antagonism Upregulates Somatostatin Receptor Subtype 2 Expression in ACTH-Producing Neuroendocrine Tumors: New Insight Based on the Selective Glucocorticoid Receptor Modulator Relacorilant. Front Endocrinol (Lausanne). 2022 Jan 4;12:793262. doi: 10.3389/fendo.2021.793262. eCollection 2021. PMID 35058882
- [Derived] Pivonello R, Bancos I, Feelders RA, Kargi AY, Kerr JM, Gordon MB, Mariash CN, Terzolo M, Ellison N, Moraitis AG. Relacorilant, a Selective Glucocorticoid Receptor Modulator, Induces Clinical Improvements in Patients With Cushing Syndrome: Results From A Prospective, Open-Label Phase 2 Study. Front Endocrinol (Lausanne). 2021 Jul 14;12:662865. doi: 10.3389/fendo.2021.662865. eCollection 2021. PMID 34335465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrolled participants who received at least 1 dose of study drug
Groups:
- Group 1: Low-dose Group: 100 mg/day for 4 weeks in Period 1, then 150 mg/day for 4 weeks in Period 2, then 200 mg/day for 4 weeks in Period 3. Period 3 was followed by a 4-week follow-up period. There was no washout between treatment periods. Per-protocol, Group 1 did not participate in Treatment Period 4.
Period: Period 1
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Started | 17 | 18
Completed | 17 | 15
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Started | 17 | 15
Completed | 16 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 3
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Started | 16 | 15
Completed | 16 | 13
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Period 4
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Started | 0 (Per-protocol, Group 1 did not participate in Period 4.) | 12 (One participant completed Period 3 but did not start Period 4 due to a pre-scheduled surgery.)
Completed | 0 | 7
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug
Groups:
- Group 1: Low-dose Group: 100 mg/day for 4 weeks in Period 1, then 150 mg/day for 4 weeks in Period 2, then 200 mg/day for 4 weeks in Period 3. Period 3 was followed by a 4-week follow-up period.
- Group 2: High-dose Group: 250 mg/day for 4 weeks in Period 1, then 300 mg/day for 4 weeks in Period 2, then 350 mg/day for 4 weeks in Period 3, then 400 mg/day for 4 weeks in Period 4. Period 4 was followed by a 4-week follow-up period.
- Total: Total of all reporting groups
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (13.62) | 49.5 (13.46) | 48.6 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 2 | 0 | 2
  Hungary | 3 | 2 | 5
  United States | 3 | 9 | 12
  Italy | 7 | 7 | 14
  United Kingdom | 2 | 0 | 2
Hypertension [Count of Participants; unit: Participants] — Confirmed with a mean systolic blood pressure (BP) of 130-170 mmHg and/or a mean diastolic BP of 85-110 mmHg based on the 24-hour ambulatory BP measurement.
  Participants | 12 | 11 | 23
Impaired Glucose Tolerance (IGT) / Type-2 Diabetes Mellitus (T2DM) [Count of Participants; unit: Participants] — Either a fasting glucose > 126 mg/dL and a 2-hour Oral Glucose Tolerance Test (oGTT) result for plasma glucose ≥ 200 mg/dL at 2 hours (for T2DM), or a 2-hour oGTT result for plasma glucose in the range of ≥ 140 mg/dL to < 200 mg/dL (for IGT).
  Participants | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Adverse Events
Description: All treatment-emergent adverse events were recorded and summarized.
Time Frame: Group 1: up to Week 16; Group 2: up to Week 20
Population: All enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Number analyzed (Participants) | 17 | 18
Participants | 15 | 18

2. Primary Outcome: Percentage of Participants With One or More Severe (≥Grade 3) Adverse Events
Description: All treatment-emergent adverse events with Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 3 (severe) were recorded and summarized.
Time Frame: Group 1: up to Week 16; Group 2: up to Week 20
Population: All enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Number analyzed (Participants) | 17 | 18
Participants | 3 | 7

3. Secondary Outcome: Percentage of Participants With Hypertension Who Experience Improvement in Blood Pressure Following Treatment With CORT125134
Description: Improvement in blood pressure was defined as a participant who experiences at least a 5 mmHg decrease in mean diastolic or systolic BP from baseline who has not taken an additional antihypertensive medication during the treatment period or increased the dosage of a concurrent antihypertensive medication.
Time Frame: Group 1: Week 12 or last observation; Group 2: Week 16 or last observation
Population: All enrolled participants with hypertension at Baseline who received at least one dose of study drug and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Number analyzed (Participants) | 12 | 11
Percentage of participants | 41.67 [15.17 to 72.33] | 63.64 [30.79 to 89.07]

4. Secondary Outcome: Percentage of Participants With IGT / T2DM Who Experienced a ≥25% Reduction in AUCglucose Following Treatment With CORT125134
Description: Improvement in glucose control was defined as a participant who experiences at least a 25% decrease from baseline in area under the concentration-time curve for blood glucose (AUCglucose) who has not taken an additional diabetes medication during the treatment period or increased the dosage of a concurrent diabetes medication.
Time Frame: Before and 0.5, 1, 1.5, and 2 hours after a glucose drink at Week 12 or last observation (Group 1) or Week 16 or last observation (Group 2)
Population: All enrolled participants with IGT / T2DM at Baseline who received at least one dose of study drug and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Number analyzed (Participants) | 13 | 14
Percentage of participants | 23.08 [5.04 to 53.81] | 0 [0 to 23.16]

5. Post Hoc Outcome: Percentage of Participants With IGT / T2DM Who Experienced Improvement in Glucose Control Following Treatment With CORT125134: Responder Definition Based on Response Criteria for Phase 3 Study NCT03697109
Description: Improvement in glucose control was defined based on response criteria for Phase 3 study NCT03697109: a participant who experiences 1) a hemoglobin A1c (HbA1c) that is decreased by ≥ 0.5% from baseline, 2) a 2-hour oGTT plasma glucose that is normalized (< 7.8 mmol/L) or decreased by ≥ 2.8 mmol/L from baseline, or 3) a total daily insulin dose that has decreased by ≥ 25% or total daily sulfonylurea dose that has decreased by ≥ 50% and an HbA1c that is unchanged or decreased from baseline.
Time Frame: as for outcome 4
Population: All enrolled participants with IGT / T2DM at Baseline who received at least one dose of study drug and had non-missing post-baseline data collected, with exclusions based on clinical judgment and/or important protocol deviations applied on a visit and outcome level rather than a participant level.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
Number analyzed (Participants) | 13 | 12
Percentage of participants | 15.38 [1.92 to 45.45] | 50.00 [21.09 to 78.91]

ADVERSE EVENTS:
Time Frame: Group 1: up to Week 16; Group 2: up to Week 20
Description: All enrolled participants who received at least 1 dose of study drug
Groups:
- Group 2: High-dose Group: 250 mg/day for 4 weeks in Period 1, then 300 mg/day for 4 weeks in Period 2, then 350 mg/day for 4 weeks in Period 3, then 400 mg/day for 4 weeks in Period 4.
Arm/Group | Group 1: Low-dose Group | Group 2: High-dose Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 4/18
Other Adverse Events (participants affected / at risk) | 15/17 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Low-dose Group (N=17) | Group 2: High-dose Group (N=18)
Pilonidal cyst (Infections and infestations) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Low-dose Group (N=17) | Group 2: High-dose Group (N=18)
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Flatulence (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Gingival hyperpigmentation (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 2
Adverse drug reaction (General disorders) | 1 | 0
Fat tissue increased (General disorders) | 1 | 0
Flushing (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 4 | 5
Pain (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 2
Application site bruise (General disorders) | 0 | 1
Application site irritation (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 5
Somnolence (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Contusion (Vascular disorders) | 1 | 0
Dizziness (General disorders) | 3 | 4
Haematoma (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Candida infection (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Application site vesicles (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Bronchitis (General disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1
Diabetes mellitus inadequate control (Endocrine disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2
Body temperature increased (Investigations) | 0 | 1
Glucocorticoids abnormal (Investigations) | 0 | 1
Drug withdrawal syndrome (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Medical device removal (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Deafness (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Astigmatism (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Polyuria (Renal and urinary disorders) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Corcept Therapeutics as the Sponsor, has a proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple Investigators and sites and Corcept Therapeutics personnel. Authorship will be established before writing of the manuscript. Because this study involves multiple centers, no individual publications will be allowed before completion of the final report of the multicenter study except as agreed with Corcept Therapeutics.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02804750/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT02804750/SAP_001.pdf